CLINICAL TRIAL: NCT01992302
Title: Risk Factors for Development of Rapid Cycling in Bipolar Disorder Patients
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Marc Valenti, MD, PhD, Hospital Clinic of Barcelona
Other Study IDs: RC-BBP
Record Dates: First submitted 2013-11-06; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Bipolar Disorder
Keywords: Rapid cycling
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Rapid Cycling Group: Patients who develop a rapid cycling course during the follow-up period.
- Non Rapid Cycling Group: Patients who do not develop a rapid cycling course during the follow-up period.

SUMMARY:
In this study we tried to elucidate the factors associated with the development of a rapid cycling course in bipolar disorder patients, in a prospective and longitudinal design, and the role of antidepressants. The identification of risk factors is extremely relevant from the clinical point of view. We hypothesized that rapid cycling bipolar disorder is associated with more chronicity, poor outcome, and more antidepressant prescription.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar I and II disorder patients according to DSM-IV criteria

Exclusion Criteria:

* Major medical comorbidities, voluntary drop-out from study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bipolar I and II disorder patients
Sampling Method: Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2004-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of patients who develop rapid cycling | 8 years

SECONDARY OUTCOMES:
Factors associated with the development of a rapid cycling course in bipolar disorder patients | 8 years

CONTACTS AND LOCATIONS:
Locations (1):
- Barcelona Bipolar Disorders Program, Hospital Clinic Barcelona, Barcelona, Catalonia, Spain